CLINICAL TRIAL: NCT04076332
Title: How "Shared Decision Making Decision-aid" Help Patients With Obstructive Sleep Apnea to Choose Treatment Plan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: N201904088
Record Dates: First submitted 2019-06-28; First posted 2019-09-03 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Shared Decision Making; OSA - Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controlled group (No Intervention): Standard oral explanation with booklet
- Decision aid group (Experimental): Shared decision making using decision aid
  Interventions: Other: Decision aid

INTERVENTIONS:
Other: Decision aid — Decision aid is a tool that helps patients become involved in decision making on choosing treatment plans. Decision aid provides information about the options and outcomes, and by clarifying personal values.
  Arms: Decision aid group

SUMMARY:
Shared decision-making helps patients to establish a treatment plan with clinicians together. Our goal was to determine if the tools we developed could reduced decisional conflict for patients with obstructive sleep apnea.

DETAILED DESCRIPTION:
Shared decision-making helps patients to establish a treatment plan with clinicians together. Our goal was to determine if the tools we developed could reduced decisional conflict for patients with obstructive sleep apnea.

Inclusion criteria: include obstructive sleep apnea patient from the outpatient clinic of Dean Wu, the sleep center of Shuang-He Hospital, 20-80 years old, polysomnography showed moderate severity (AHI ≥ 15), can communicate in Chinese.

Exclusion criteria: dementia, mental illness, language difficulties.

ELIGIBILITY:
Inclusion Criteria:

* Include obstructive sleep apnea patient from the outpatient clinic of Dean Wu, the sleep center of Shuang-He Hospital, 20-80 years old, polysomnography showed moderate severity (AHI ≥ 15), can communicate in Chinese

Exclusion Criteria:

* Exclude dementia, mental illness, language difficulties

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Decision conflict | Immediately after patient received standard oral explanation with booklet or decision aids at out-patient department
  We'd like to measure the score of SURE test, which published by Légaré at 2008, as a decisional conflict scale. SURE includes 4 questions representing "sure of myself, understand information, risk-benefit ratio, encouragement". Each question consisted of a typical five-level Likert item (strongly disagree, disagree, neither agree nor disagree, agree, strongly agree).

SECONDARY OUTCOMES:
Health literacy | Immediately after patient received standard oral explanation with booklet or decision aids at out-patient department
  Self-evaluation score of health literacy. We measure health literacy via one question of SURE test (Sure of myself - Do you feel SURE about the best choice for you?). This question also consisted of a typical five-level Likert item (strongly disagree, disagree, neither agree nor disagree, agree, strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Dean Wu, MD, PhD, Study Chair — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kapur VK, Auckley DH, Chowdhuri S, Kuhlmann DC, Mehra R, Ramar K, Harrod CG. Clinical Practice Guideline for Diagnostic Testing for Adult Obstructive Sleep Apnea: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2017 Mar 15;13(3):479-504. doi: 10.5664/jcsm.6506. PMID 28162150
- [Result] Epstein LJ, Kristo D, Strollo PJ Jr, Friedman N, Malhotra A, Patil SP, Ramar K, Rogers R, Schwab RJ, Weaver EM, Weinstein MD; Adult Obstructive Sleep Apnea Task Force of the American Academy of Sleep Medicine. Clinical guideline for the evaluation, management and long-term care of obstructive sleep apnea in adults. J Clin Sleep Med. 2009 Jun 15;5(3):263-76. PMID 19960649
- See also: American Academy of Sleep Medicine Practice Guidelines — https://aasm.org/clinical-resources/practice-standards/practice-guidelines/
- See also: UpToDate: Obstructive sleep apnea and cardiovascular disease in adults — https://www.uptodate.com/contents/obstructive-sleep-apnea-and-cardiovascular-disease-in-adults
- See also: UpToDate: Sleep-related breathing disorders and stroke — https://www.uptodate.com/contents/sleep-related-breathing-disorders-and-stroke